CLINICAL TRIAL: NCT03393143
Title: PCORI-1609-36568 A Naturalistic Experiment Evaluating the Impact of Medicaid Treatment Reimbursement Changes on Opioid Prescribing and Patient Outcomes Among Patients With Back Pain
Brief Title: A Naturalistic Experiment Evaluating the Impact of Medicaid Treatment Reimbursement Changes on Opioid Prescribing and Patient Outcomes Among Patients With Back Pain
Acronym: Back on Track
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); OCHIN, Inc. (Other); Harvard Pilgrim Health Care (Other)
Responsible Party: Sponsor
Other Study IDs: R217083
Record Dates: First submitted 2017-12-27; First posted 2018-01-08 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Back Pain; Neck Pain
Keywords: Primary Health Care; Analgesics, Opioid; Medicaid
MeSH Terms: conditions — Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oregon patients: Adult Medicaid patients with back pain who get their care in community health clinics in Oregon
- California patients: Adult Medicaid patients with back pain who get their care in community health clinics in California

SUMMARY:
Back on Track is a quasi-experimental, mixed-methods study of a unique natural experiment that will answer the question: what is the comparative effectiveness of different payer or health-system strategies that aim to prevent unsafe opioid prescribing? The State of Oregon is enacting a Medicaid reimbursement policy to enhance access to evidence-based non-pharmacotherapeutic treatment options while restricting reimbursement for opioids for back pain. We will assess whether the policy decreases unsafe opioid prescribing and improves patient outcomes compared with usual back pain treatment practices in a comparable state, California, that is not changing Medicaid payment policy.

DETAILED DESCRIPTION:
Back pain is one of the most common reasons patients seek medical care, and it can have a big impact on patients' quality of life and functioning. Patients and providers are becoming more frustrated with common back pain treatments like the long-term use of opioid medications and steroid injections, which have been shown to have limited long-term impact on patients' pain and day-to-day functioning and can have safety risks.

The State of Oregon recently changed what back and neck pain treatments they cover for its Medicaid enrollees. This started to affect those insured by Medicaid in July 2016 and was implemented by January 2018. These changes ended payments for treatments like long-term opioid therapy and injections. They also expanded coverage for nondrug treatments, such as acupuncture, osteopathic or chiropractic manipulation, physical/occupational therapy, and cognitive behavioral therapy. While experts agree that opioid use must be reduced, Oregon is among the first states to try such strong measures to promote nondrug treatments and prevent the use of long-term opioid treatment for back and neck pain.

The Oregon Medicaid reimbursement changes for back and neck pain treatment create the opportunity for a "natural experiment." In this mixed-methods, observational study, we will evaluate the impact of the reimbursement changes by comparing outcomes among patients with back pain in Oregon who will have access to these expanded nondrug treatments to similar patients seen in comparable clinics in California where expanded services for back and neck pain are not covered by the type of comprehensive payer incentive undertaken in Oregon.

Specifically, we will use electronic health record, Medicaid claims data, and data obtained from a longitudinal patient survey to assess the impact of the changes on:

* Patients' pain severity, pain related functioning, and satisfaction with care
* Patients' use of pain-related health care services
* Opioid use
* Unintended consequences, such as the use of illicit drugs (While we expect the Oregon Medicaid change to result in many positive changes, limiting the use of opioids and pain reducing procedures like injections may motivate some individuals to use drugs that were not prescribed by their doctor.)

In addition, we will use qualitative research methods to characterize the facilitators and barriers experienced by patients, health care providers, and clinic administrators and staff in adopting the Medicaid reimbursement changes and their satisfaction with the constellation of available and utilized services.

Thus, this study has three components: 1) patient survey, 2) administrative data-based study (data-only), and 3) qualitative evaluation. This record focuses on the component of the study in which subjects are able to enroll - the patient survey.

ELIGIBILITY:
Inclusion criteria:

1. Adults age 18-65 years
2. Insured by Medicaid
3. Have back or neck pain (based on ICD-CM diagnosis)
4. Receive their primary health care at participating OCHIN member federally qualified health centers in Oregon and California

Exclusion criteria:

1. Patients with current malignant cancer diagnosis
2. Any evidence of patient having received hospice or other end-of-life palliative care within the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient survey: Medicaid-insured adults age 18-65 years who are diagnosed with back or neck pain and receive their primary health care from participating OCHIN member federally-qualified health centers in Oregon and California. Patients may have acute or chronic pain and may be receiving long-term opioid therapy or not receiving long-term opioid therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2748 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Pain severity | Baseline to 12 months
  Modified 10-item version of the Brief Pain Inventory-Short Form (BPI-SF), composite of pain intensity (3 items) and pain-related interference (7 items) subscales (10 items total; continuous)
Use of pain-related services | Baseline to 12 months
  Use of pain-related services will be assessed by asking about use (Yes/no; binary) of the following pain-related services: Acupuncture, Chiropractic, Massage Therapy, Rehabilitation Therapies; Cognitive Behavioral Therapy (CBT) or Acceptance and Commitment Therapy (ACT); Psychotherapy, Yoga Group or Class, and Stretching/Strengthening Exercise Therapy.
Patient satisfaction with health care services | Baseline to 12 months
  Patient satisfaction with health care services will be assessed by asking the following question:
  How satisfied have you been with the services you've received to help you manage your pain? (0-10 scale; continuous; higher score = more satisfied)
Negative outcomes related to pain services | Baseline to 12 months
  Negative outcomes related to pain services will be assessed by asking the following question: Have you had any problems or bad outcomes from services that you have received or things you've done to manage your pain? (Yes/no; binary) If respond yes, a description of the problem or bad outcome is collected.
Illicit drug use | Baseline to 12 months
  Illicit drug use will be assessed by asking the following four questions:
  Have you used an opioid prescription medication that was not prescribed for you by your health care provider? (Yes/no; binary)
  Have you used any street drugs to manage your pain? (Yes/no; binary) If respond yes, a description of the street drug(s) is collected.
  Have you used any other types of prescription medications that were not prescribed for you by a health care provider to manage your pain? (Yes/no; binary) If respond yes, a description of the prescription medication(s) is collected.
  Have you used heroin to manage your pain? (Yes/no; binary)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn DeBar, PhD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- OCHIN, Inc., Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No